CLINICAL TRIAL: NCT04186676
Title: Myocardial Infarction With Non-Obstructive Coronary Arteries in the Greek Population: Diagnosis and Management (The MINOCA-GR Registry)
Brief Title: Myocardial Infarction With Non-Obstructive Coronary Arteries in the Greek Population
Acronym: MINOCA-GR
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: New York University (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, George Giannakoulas, Associate Professor, MD, PhD, AHEPA University Hospital
Other Study IDs: CIP_001_MINOCA_GR_27.11.2019
Record Dates: First submitted 2019-11-29; First posted 2019-12-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Acute Myocardial Infarction; Non-Obstructive Coronary Atherosclerosis; Ischemic Heart Disease; Angina Pectoris; Coronary Microvascular Disease
Keywords: MINOCA; Myocardial Infarction; Cardiac Computed Tomography Angiography; Angina; Leiden CTA risk score; Indexed Coronary Volume
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Microvascular Angina; MINOCA; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MINOCA patients: Prevalence, demographics, clinical profile, previous anginal status, presence of cardiovascular risk factors, management and outcomes in consecutive patients with Myocardial Infarction with Non-Obstructive Coronary Arteries admitted to study clinical sites
  Interventions: Other: MINOCA registry; Diagnostic Test: CCTA Phenotypes

INTERVENTIONS:
Other: MINOCA registry — Prevalence, demographics, clinical profile, anginal status, presence of cardiovascular risk factors, management and outcomes
Diagnostic Test: CCTA Phenotypes — 1. Complete normal coronary arteries
  2. Diffuse non-obstructive coronary artery disease
  3. Non-obstructive high-risk plaques
  4. Myocardial bridges

SUMMARY:
The MINOCA-GR registry will be the first nationwide study aiming to obtain data regarding prevalence, demographics, clinical profile, previous anginal status, presence of cardiovascular risk factors, management and outcomes in patients with Myocardial Infarction with Non-Obstructive Coronary Arteries. An additional purpose of the registry is to highlight, for the first time worldwide to the best of the investigator's knowledge, the role of cardiac computed tomography angiography for risk stratification and personalized therapeutic approach in MINOCA patients.

DETAILED DESCRIPTION:
MINOCA occurs in 5%-10% of all patients with Acute Myocardial Infarction (AMI) and these patients are younger and more often women in comparison with patients with AMI and obstructive Coronary Artery Disease (CAD). The underlying pathophysiological mechanisms are poorly understood, although several different mechanisms have been proposed, including plaque disruption, spasm, thromboembolism, dissection, microvascular dysfunction and ischemic myocardial injury attributable to supply/demand mismatch. In most, but not all, studies of prognosis, MINOCA patients had better outcomes than their AMI counterparts with coronary artery disease but faced a high risk for recurrent events, with one study finding that 25% of patients with MINOCA experience angina in the following year. Optimal patient management requires early diagnosis as well as understanding which of the myriad of mechanisms (atherosclerotic or non-atherosclerotic as well as a combination of both) may be underlying the initial diagnosis. The effects of secondary preventive treatments proven beneficial in patients with classical type I AMI are unknown in MINOCA patients; randomized clinical trials, and large observational studies, as well, evaluating different treatments in MINOCA patients do not exist. Hence, evidence-based guidelines for treatment of MINOCA are lacking. Elucidating the associations between different treatments and outcome may also increase the understanding of underlying mechanisms of MINOCA. The underlying mechanisms strongly determine prognosis and more importantly, therapeutic interventions as well as their success.

Likewise, multimodality imaging could provide new insights into the management of MINOCA patients. The current research reveals the utility of Cardiac Magnetic Resonance for diagnosis and risk stratification of suspected MINOCA patients but at the same time shows how much more information is needed to further characterize risk and ultimately develop therapeutic approaches to alter its natural history. Computed tomography has a suite of strengths including diagnosis of CAD, identification of plaque characteristics, morphology and perfusion data, and even possibly delayed enhancement; its ability to detect nonobstructive coronary disease by way of visualizing not only the lumen but also plaques is very helpful in our efforts trying to understand microvascular disease, plaque erosion, and myocardial infarction with no obstructive coronary artery. Furthermore, up until recently, high-risk plaque features and lesion specific ischemia are thought to be not directly related. However, emerging evidence suggests a possible relationship between high-risk plaque features, particularly low attenuation plaque volume and positive remodeling, with lesion specific ischemia by fractional flow reserve. Such relationship is independent of degree of luminal stenosis. As a result of the above, it is obvious that Cardiac Computed Tomography Angiography (CCTA) may have a potential role in some selected patients with MINOCA, depending on their clinical picture and stability.

Regarding Greece, the MINOCA-GR registry will be the first prospectively enrolling medical database of this magnitude.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Patients without known history of coronary artery disease
3. Patients with acute coronary syndrome with and/or without ST-segment elevation who underwent coronary angiography within 24h after onset of the disease
4. Absence of obstructive coronary atherosclerosis (normal coronary arteries or plaques <50% stenosis) based on the results of invasive coronary angiography
5. Subject has provided written informed consent
6. Subject is willing to comply with study follow-up requirements

Exclusion Criteria:

1. Patients < 18 years old at time of coronary angiography
2. Patients with a previous history of coronary artery disease and/or prior revascularization
3. Patients with serious concurrent disease and life expectancy of < 1 year
4. Patients who refuse to give written consent for participation in the study
5. In the investigator's opinion, subject will not be able to comply with the follow-up requirements
6. Subject is pregnant and/or breastfeeding or intends to become pregnant during the study
7. Subject has a known allergy to contrast agent that cannot be adequately pre-medicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll consecutive patients with MINOCA admitted to study clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Frequency of post-MI angina [Seattle Angina Questionnaire (SAQ)] | 1 month
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life).
Frequency of post-MI angina [Seattle Angina Questionnaire (SAQ)] | 6 months
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life).
Frequency of post-MI angina [Seattle Angina Questionnaire (SAQ)] | 12 months
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life).
Extent of coronary atherosclerosis | 15 days after the acute event
  Total atherosclerotic plaque volume (mm3)
Extent of coronary atherosclerosis using Leiden CTA risk score | 15 days after the acute event
  Leiden CTA risk score incorporates the presence, extent, severity, location, and composition of coronary artery disease (CAD). Leiden CTA score is calculated using the following approach. First, the presence of CAD is determined in each segment. When plaque is absent the score is 0. When plaque is present a score of 1.1, 1.2 or 1.3 is given according to plaque composition (calcified, noncalcified, and mixed plaque, respectively). Subsequently, this score is multiplied by a weight factor for the location of the segment in the coronary artery tree (0.5 through 6 according to vessel, proximal location and system dominance) and multiplied by a weight factor for stenosis severity (1.4 for ≥50% stenosis and 1.0 for stenosis <50%). The final score (range 0 to 42) is calculated by addition of the individual segment scores. Leiden CTA risk score calculator is available at: http://18.224.14.19/calcApp/.
Extent of coronary atherosclerosis using Gensini score | 15 days after the acute event
  The relative severity of a lesion is indicated using a score of 1 for 1-25% obstruction and doubling that number as the severity of obstruction progresses with each step in the 25-50-75-90-99-100% diameter reduction. Thus, the severity score for each lesion may range from 1 to 32. Furthermore, the score weighed according to the usual blood flow to the left ventricle in each vessel or vessel segment. A multiplying factor is applied to each lesion score based upon its location in the coronary tree, depending on the functional significance of the area supplied by that segment. If a segment is totally occluded or 99% stenosed and receiving collaterals, a collateral adjustment factor is used, and the adjustment is reduced by the extent of disease in the vessel that is the source of collaterals. The final score is the sum of all the lesion scores (Reference: Rampidis GP et al. A guide for Gensini Score calculation. Atherosclerosis 2019 August 2019;287:181-183).

SECONDARY OUTCOMES:
Indexed Coronary Volume | 15 days after the acute event
  Calculated by dividing the total coronary volume to the left ventricle (LV) mass, both derived from CCTA (mm3/gr)
Generic health status [Medical Outcomes Study 12-Item Short Form (SF-12)] | 12 months
  The Medical Outcomes Study 12-Item Short Form (SF-12) is a general health questionnaire and is computed using the scores of 12 questions ranging from 0 to 100, where 0 indicates the lowest level of health and 100 indicates the highest level of health.
Chest-pain rehospitalization | 12 months
  Frequency (%) of chest-pain rehospitalization
Hospitalization for a bleeding event | 12 months
  Frequency (%) of hospitalization for a bleeding event
Frequency of occurrence of high-risk plaques | 15 days after the acute event
  Frequency (%) of occurrence of high-risk plaque features (HU <30, remodelling index > 1.1, napkin-ring sign, spotty calcium)
Atrial Fibrillation | 12 months
  Frequency (%) of occurrence of atrial fibrillation
Heart Failure | 12 months
  Frequency (%) of occurrence of acute decompensated heart failure with or without cardiogenic shock

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Giannakoulas, MD, PhD, Principal Investigator — AHEPA University Hospital of Thessaloniki
Locations (3):
- Greece (3):
  - General Hospital of Veroia, Véroia, Imathia
  - National & Kapodistrian University of Athens, First Department of Cardiology, Hippokration Hospital, Athens
  - AHEPA University Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rampidis GP, Benetos G, Benz DC, Giannopoulos AA, Buechel RR. A guide for Gensini Score calculation. Atherosclerosis. 2019 Aug;287:181-183. doi: 10.1016/j.atherosclerosis.2019.05.012. Epub 2019 May 10. No abstract available. PMID 31104809
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Tamis-Holland JE, Jneid H, Reynolds HR, Agewall S, Brilakis ES, Brown TM, Lerman A, Cushman M, Kumbhani DJ, Arslanian-Engoren C, Bolger AF, Beltrame JF; American Heart Association Interventional Cardiovascular Care Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; and Council on Quality of Care and Outcomes Research. Contemporary Diagnosis and Management of Patients With Myocardial Infarction in the Absence of Obstructive Coronary Artery Disease: A Scientific Statement From the American Heart Association. Circulation. 2019 Apr 30;139(18):e891-e908. doi: 10.1161/CIR.0000000000000670. PMID 30913893
- [Background] Grodzinsky A, Arnold SV, Gosch K, Spertus JA, Foody JM, Beltrame J, Maddox TM, Parashar S, Kosiborod M. Angina Frequency After Acute Myocardial Infarction In Patients Without Obstructive Coronary Artery Disease. Eur Heart J Qual Care Clin Outcomes. 2015;1(2):92-99. doi: 10.1093/ehjqcco/qcv014. Epub 2015 Jul 23. PMID 28239487
- [Background] Ahmadi A, Leipsic J, Ovrehus KA, Gaur S, Bagiella E, Ko B, Dey D, LaRocca G, Jensen JM, Botker HE, Achenbach S, De Bruyne B, Norgaard BL, Narula J. Lesion-Specific and Vessel-Related Determinants of Fractional Flow Reserve Beyond Coronary Artery Stenosis. JACC Cardiovasc Imaging. 2018 Apr;11(4):521-530. doi: 10.1016/j.jcmg.2017.11.020. Epub 2018 Jan 5. PMID 29311033
- [Background] Nordenskjold AM, Lagerqvist B, Baron T, Jernberg T, Hadziosmanovic N, Reynolds HR, Tornvall P, Lindahl B. Reinfarction in Patients with Myocardial Infarction with Nonobstructive Coronary Arteries (MINOCA): Coronary Findings and Prognosis. Am J Med. 2019 Mar;132(3):335-346. doi: 10.1016/j.amjmed.2018.10.007. Epub 2018 Oct 25. PMID 30367850
- [Background] van Rosendael AR, Shaw LJ, Xie JX, Dimitriu-Leen AC, Smit JM, Scholte AJ, van Werkhoven JM, Callister TQ, DeLago A, Berman DS, Hadamitzky M, Hausleiter J, Al-Mallah MH, Budoff MJ, Kaufmann PA, Raff G, Chinnaiyan K, Cademartiri F, Maffei E, Villines TC, Kim YJ, Feuchtner G, Lin FY, Jones EC, Pontone G, Andreini D, Marques H, Rubinshtein R, Achenbach S, Dunning A, Gomez M, Hindoyan N, Gransar H, Leipsic J, Narula J, Min JK, Bax JJ. Superior Risk Stratification With Coronary Computed Tomography Angiography Using a Comprehensive Atherosclerotic Risk Score. JACC Cardiovasc Imaging. 2019 Oct;12(10):1987-1997. doi: 10.1016/j.jcmg.2018.10.024. Epub 2019 Jan 16. PMID 30660516
- [Background] Benetos G, Buechel RR, Goncalves M, Benz DC, von Felten E, Rampidis GP, Clerc OF, Messerli M, Giannopoulos AA, Gebhard C, Fuchs TA, Pazhenkottil AP, Kaufmann PA, Grani C. Coronary artery volume index: a novel CCTA-derived predictor for cardiovascular events. Int J Cardiovasc Imaging. 2020 Apr;36(4):713-722. doi: 10.1007/s10554-019-01750-2. Epub 2020 Jan 1. PMID 31894527
- [Background] Benz DC, Benetos G, Rampidis G, von Felten E, Bakula A, Sustar A, Kudura K, Messerli M, Fuchs TA, Gebhard C, Pazhenkottil AP, Kaufmann PA, Buechel RR. Validation of deep-learning image reconstruction for coronary computed tomography angiography: Impact on noise, image quality and diagnostic accuracy. J Cardiovasc Comput Tomogr. 2020 Sep-Oct;14(5):444-451. doi: 10.1016/j.jcct.2020.01.002. Epub 2020 Jan 13. PMID 31974008
- [Derived] Rampidis GP, Kampaktsis PNu, Kouskouras K, Samaras A, Benetos G, Giannopoulos AAlpha, Karamitsos T, Kallifatidis A, Samaras A, Vogiatzis I, Hadjimiltiades S, Ziakas A, Buechel RR, Gebhard C, Smilowitz NR, Toutouzas K, Tsioufis K, Prassopoulos P, Karvounis H, Reynolds H, Giannakoulas G. Role of cardiac CT in the diagnostic evaluation and risk stratification of patients with myocardial infarction and non-obstructive coronary arteries (MINOCA): rationale and design of the MINOCA-GR study. BMJ Open. 2022 Feb 2;12(2):e054698. doi: 10.1136/bmjopen-2021-054698. PMID 35110321